CLINICAL TRIAL: NCT06738862
Title: [18F] - FD17 PET Imaging of α-synuclein: A Clinical Study in α-synucleinopathy Patients
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: [18F]-FD17 PET
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: α-synucleinopathy; Parkinson's Disease (PD); Multiple System Atrophy; Rapid Eye Movement Sleep Behavior Disorder; PET
MeSH Terms: conditions — Multiple System Atrophy; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- PD group
  Interventions: Other: PET
- MSA group
  Interventions: Other: PET
- RBD group
  Interventions: Other: PET
- HC group
  Interventions: Other: PET

INTERVENTIONS:
Other: PET — [18F] - FD17 PET imaging

SUMMARY:
The main objective of this study is to establish a standardized method for [18F] - FD17 PET imaging in α-synucleinopathy patients, and to analyze its physiological distribution in healthy individuals as well as its pathological distribution in α-synucleinopathy patients, including Parkinson's disease (PD), multiple system atrophy (MSA), and idiopathic rapid-eye-movement sleep behavior disorder (iRBD). Specifically, [18F] - FD17 PET imaging focuses on evaluating the deposition of α-synuclein and exploring the diagnostic value of [18F] - FD17 PET in PD, MSA, and iRBD patients. In addition, for PD, MSA and RBD patients, dopamine transporter(DAT)-PET imaging was performed to evaluate the distribution and density of DAT in brain. The study aims not only to clarify the specific binding mode of the imaging agent in different α-synucleinopathies, but also to evaluate its efficacy and potential application prospects in early diagnosis , providing new methods for the diagnosis and treatment of neurodegenerative diseases. This study is expected to contribute to early pathological detection and accurate diagnosis in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 1: Normal cognitive function, CDR score=0（for healthy subjects）

  2: Without neurological disorders, major chronic diseases, malignant tumors, or acute infectious diseases (for healthy subjects）

  3: Without the family history of neurological disorders related to motor or cognitive impairments(for healthy subjects）

  4: Clinical diagnosis of idiopathic PD (for PD patients)

  5: Clinical diagnosis of MSA (for MSA patients)

  6: Clinical diagnosis of idiopathic RBD (for RBD patients)

  7: An informed consent form signed in writing by the subject or their legal guardian or caregiver.

  8: Must be abled to be accompanied by nursing staff

  9: Must be able to understand and sign a informed consent form before any evaluation and examination

  10: Must have medical records to prove that they have undergone surgical sterilization (such as hysterectomy, bilateral oophorectomy, or tubal ligation) or menopause for more than one year.(for female subjects)

  11: Must adopt isolation contraception measures within 3 months after the start of this study.(for female subjects)

  12: Willing and capable to cooperate with all projects of this study.

Exclusion Criteria:

* 1: Other severe neurological disorders. Gastrointestinal, cardiovascular, liver, kidney, hematological, tumor, endocrine, respiratory, immunodeficiency, and other serious diseases.

  2: Received ionizing radiation outside the scope of this experiment, resulting in an annual radiation exposure dose exceeding 50 mSv in the past year,

  3: History of drug abuse or alcoholism

  4: Pregnant or lactating women

  5: Poor venous conditions, unable to tolerate repeated venipuncture

  6: Received experimental drug or device treatment with unclear efficacy or safety in last 1 month.

  7: Any situation that the investigators believe may cause harm or potential harm in any aspect related to this study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 PD subjects ,10 MSA subjects, 10 RBD subjects ,and 5 healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-12-14 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
electrocardiogram | 2 weeks ahead of and after [18F] - FD17 PET/MRI
  Heart rate, atrial rate, ventricular rate, P-R interval, QRS axis, QRS duration, QRS potential, and all other electrocardiographic indicators will be collected by 12-lead electrocardiogram. These outcomes will be used to figure out whether the subjects have a potential heart disease and whether [18F] - FD17 PET/MRI will do harm to subjects.
routine blood test | 2 weeks ahead of and after [18F] - FD17 PET/MRI
  10ml peripheral venous blood will be collected and to measure red blood cell cell count and percentage, hemoglobin content, white blood cell count and percentage, platelet count, and all other indicators in routine blood test. These outcomes will be used to figure out whether the subjects have a potential disease and whether [18F] - FD17 PET/MRI will do harm to subjects.
routine urine test | 2 weeks ahead of and after [18F] - FD17 PET/MRI
  20ml urine will be collected for routine urine test. Indicators including red blood cell and white blood cell count under a microscope, urine specific gravity, urine PH, urinary protein, glucose in urine and all others will be measured. These outcomes will be used to figure out whether the subjects have a potential disease and whether [18F] - FD17 PET/MRI will do harm to subjects.
liver renal function test | 2 weeks ahead of and after [18F] - FD17 PET/MRI
  10ml peripheral venous blood will be collected and to measure alanine aminotransferase(ALT), aspartate aminotransferase(AST), alkaline phosphatase(ALP), Gamma-glutamyltransferase(GGT), creatinine, urea nitrogen, uric acid and all other liver renal function test indicators in serum. These outcomes will be used to figure out whether the subjects have potential hepatorenal dysfunction and whether [18F] - FD17 PET/MRI will do harm to subjects.

SECONDARY OUTCOMES:
[18F] - FD17 PET imaging results | Baseline

OTHER OUTCOMES:
DAT(dopamine transporter) PET imaging results | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of neurology, Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No